CLINICAL TRIAL: NCT01059188
Title: Preoperative Chemotherapy and Radiotherapy Concomitant to Cetuximab in Non-Small Cell Lung Cancer (NSCLC) Patients With IIIB Disease - A Multicenter Phase II Trial
Brief Title: Neo-adjuvant Treatment in Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 16/08; SWS-SAKK-16/08; EU-21002; CDR0000664070
Record Dates: First submitted 2010-01-28; First posted 2010-01-29 (Estimated); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; adenocarcinoma of the lung; adenosquamous cell lung cancer; large cell lung cancer; squamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Cetuximab; Cisplatin; Docetaxel; Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cetuximab, Cisplatin, Docetaxel, Radiotherapy and Surgery (Experimental)
  Interventions: Drug: cetuximab; Drug: cisplatin; Drug: docetaxel; Radiation: Radiotherapy; Procedure: Surgery

INTERVENTIONS:
Drug: cetuximab — 400 mg/m2 initial dose on day 1 250 mg/m2 weekly starting on day 8 and for 12 weeks
  Other Names: Erbitux
Drug: cisplatin — 50 mg/m2 on day 1 and 2 of 21 day cycles, for 3 cycles
  Other Names: Platin
Drug: docetaxel — 85 mg/m2 day 1 of 21 day cycles, for 3 cycles
  Other Names: Taxotere
Radiation: Radiotherapy — 44 Gy (PTV1=30 Gy, PTV2=14 Gy), for 3 weeks, after the 3 cycles of Cisplatin / Docetaxel treatment
Procedure: Surgery — Ipsilateral formal mediastinal lymphadenectomy. In case of involved N3 lymph nodes, resection of the precarinal and contralateral nodes.

SUMMARY:
RATIONALE: Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as cisplatin and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Giving these treatments before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase II trial is studying the side effects of giving cetuximab together with cisplatin and docetaxel before radiation therapy and cetuximab followed by surgery and to see how well it works in treating patients with stage IIIB non-small cell lung cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the efficacy and safety of neoadjuvant sequential chemoimmunotherapy comprising cetuximab, cisplatin, and docetaxel before radiotherapy and cetuximab followed by surgery in patients with resectable stage IIIB non-small cell lung cancer.

OUTLINE: This is a multicenter study.

* Chemoimmunotherapy (courses 1-3): Patients receive chemoimmunotherapy comprising cetuximab IV over 1-2 hours on days 1, 8, and 15; cisplatin IV over 1 hour on days 1 and 2; and docetaxel IV over 1 hour on day 1. Patients also receive filgrastim (G-CSF) on days 3-8 or a single dose of pegfilgrastim the day after chemotherapy. Treatment repeats every 3 weeks for 3 courses.
* Radiotherapy (course 4): Beginning on day 1 of week 10, patients undergo 3-dimensional conformal or intensity-modulated radiotherapy 5 days a week for 3 weeks. Patients also receive cetuximab IV over 1 hour on days 1, 8, and 15.
* Surgery: Beginning 21-28 days after completion of radiotherapy, patients undergo surgery.

After completion of study treatment, patients are followed every 3 months for 2 years and every 6 months for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell lung cancer (NSCLC)

  * Squamous, adeno, large cell, or poorly differentiated disease
  * Stage IIIB disease (T4N0-3M0 or T1-4N3M0) according to 6th TNM classification

    * Assessed by bronchoscopy and PET-CT scan within 42 days of registration
    * No malignant pleural or pericardial effusion, invasion of the aorta, esophagus, myocardium, or supraclavicular
    * No scalene nodes N3
    * No stages IIIB disease defined only by satellite lesions in the same lobe
* Lymph node staging done by mediastinoscopy (or EBUS) in N+ disease on PET-CT scan (SUV above mediastinum background SUV) or CT (size > 10 mm in the smallest diameter) within 42 days of registration

  * Fine needle aspiration biopsy must be done by EBUS, TBNA, or VATS if lymph nodes are not accessible by mediastinoscopy (ATS nodes #5/6)
  * Mediastinoscopy is mandatory for suspicion of T4 tumor invading the trachea on PET-CT and CT scan in N-disease
* Measurable disease assessed by contrast-enhanced CT-scan within 28 days of registration
* Tumor tissue available for translational research (no cytology)
* Resectable disease based on a multidisciplinary tumor board decision
* No brain metastasis (confirmed by MRI within 42 days of registration)

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Platelet count ≥ 100 x 10^9/L
* Neutrophil count ≥ 1.5 x 10^9/L
* Bilirubin normal
* AST ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* Creatinine clearance ≥ 60 mL/min
* FEV1 and DLCO ≥ 80% OR exercise test peak V02 > 75% or 20 mL kg^-1 min^-1 (for pneumonectomy)
* Exercise test peak V02 ≥ 35% and ≥ 10 mL kg^-1 min^-1 with predicted postoperative FEV1 and DLCO ≥ 30% (for resection less than pneumonectomy [resection up to calculated extend according to ESTS/ACCP guidelines])
* Ejection fraction > 45% assessed by echocardiography
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 months after completion of study therapy
* Must be compliant and geographically proximal for proper staging and follow-up
* No previous malignancy within the past 5 years except for adequately treated carcinoma in situ of the cervix or localized nonmelanoma skin cancer
* No psychiatric disorder precluding understanding of information on trial-related topics and giving informed consent
* No preexisting peripheral neuropathy > grade 1
* No ischemia or relevant dysfunction revealed by noninvasive stress testing (stress radionuclide myocardial perfusion imaging or dobutamine stress echocardiography) for patients with a history of ischemic heart disease or any other relevant cardiovascular condition
* No unstable cardiac disease requiring treatment, congestive heart failure or angina pectoris even if medically controlled, significant arrhythmia, or myocardial infarction within the past 3 months
* No serious underlying medical condition that, at the judgment of the investigator, could impair the ability of the patient to participate in the trial (e.g., active autoimmune disease, uncontrolled diabetes, or uncontrolled infection)
* No known hypersensitivity to trial drugs or hypersensitivity to any other component of the trial drugs
* No absolute contraindications for the use of corticosteroids as premedication

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy to the chest
* No pretreatment with any cytostatic therapy
* No concurrent corticosteroids, except for prophylactic medication regimen prior to treatment or treatment of acute hypersensitivity reactions or chronic treatment (initiated > 6 months prior to trial entry) at low-dose (< 20 mg methylprednisolone or equivalent)
* No concurrent drugs contraindicated for use with the trial drugs
* At least 30 days since prior and no other concurrent experimental drugs or other anticancer therapy on another clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2010-05-03 (Actual); Primary Completion 2016-12-09 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | at 1 year (+/- 1 month)

SECONDARY OUTCOMES:
Treatment-related death during chemoimmunotherapy, radioimmunotherapy, and perioperatively | 30 days after surgery
Metabolic response evaluated by PET | At baseline and after chemo-immunotherapy
Response status after chemoimmunotherapy and radioimmunotherapy | After chemoimmunotherapy and after radioimmunotherapy
Complete pathological response | After surgery
Overall survival | At the end of the follow-up phase (max. 5 years after treatment termination or surgery)
Adverse events | During the all trial treatment until 30 days after surgery or treatment stop
Operability | Before trial treatment

CONTACTS AND LOCATIONS:
Overall Officials: Solange Peters, MD, Study Chair — Centre Hospitalier Universitaire Vaudois; Daniel C. Betticher, MD, Study Chair — Kantonsspital Freiburg; Miklos Pless, Prof, Study Chair — Kantonsspital Winterthur KSW; Roger Stupp, MD, Study Chair — Centre Hospitalier Universitaire Vaudois
Locations (15):
- Switzerland (15):
  - Saint Claraspital AG, Basel
  - Universitaetsspital-Basel, Basel
  - Istituto Oncologico della Svizzera Italiana - Ospedale San Giovanni, Bellinzona
  - Inselspital Bern, Bern
  - Spitalzentrum Biel, Biel
  - Kantonsspital Bruderholz, Bruderholz
  - Kantonsspital Graubuenden, Chur
  - Hopital Fribourgeois, Fribourg
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Liestal, Liestal
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Regionalspital, Thun
  - Kantonsspital Winterthur, Winterthur
  - UniversitaetsSpital Zuerich, Zurich

IPD SHARING:
Plan to Share IPD: No